CLINICAL TRIAL: NCT02738749
Title: Sodium Channel Splicing in Heart Failure Trial (SOCS-HEFT) Prospective Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rhode Island Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 426228-16
Record Dates: First submitted 2016-04-07; First posted 2016-04-14 (Estimated); Last update posted 2017-04-12 (Actual); Status verified 2017-04

CONDITIONS: Death, Sudden, Cardiac
Keywords: sudden cardiac death, sodium channel splicing variant
MeSH Terms: conditions — Death, Sudden, Cardiac | interventions — Defibrillators, Implantable

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ICD group (Other): Adult patients with newly implanted ICD devices for primary prevention will be enrolled. At baseline, 3-, 6-, 9-, and 12-month followup visit, the medial information and blood samples will be collected.
  Interventions: Device: Implantable cardioverter-defibrillator (ICD)

INTERVENTIONS:
Device: Implantable cardioverter-defibrillator (ICD) — Patients with newly implanted implantable cardioverter-defibrillators (ICDs) for primary prevention will be enrolled.

SUMMARY:
Congestive heart failure (CHF) represents a major health care concern in the United States. Currently, risk stratification of sudden cardiac death and the need for implantable cardioverter-defibrillator (ICD) placement are essentially dependent upon assessment of left ventricular ejection fraction (LVEF). Nevertheless, the predictive value of LVEF is suboptimal, alternative testing for risk assessment for the development of sudden cardiac death in the heart failure population is desirable.

At the genome level, the investigator has focused on the role of SCN5A gene mutations in arrhythmogenesis. Lymphocyte SCN5A mRNA processing may serve as a surrogate marker to assess SCN5A function at the cardiac level and may correlated with arrhythmic risk in high risk populations. This study will determine if SCN5A variant levels are predictive of appropriate ICD therapies in patients with a newly implanted ICD.

DETAILED DESCRIPTION:
Scientific Background and Significance Introduction

Congestive heart failure (CHF) represents a major health care concern in the United States. It has been estimated that approximately 5 million patients in the U.S. have CHF, and nearly 550,000 people are diagnosed with this disease annually. It is known that sudden cardiac death occurs more frequently in the setting of structural heart disease. Moreover, the risk for sudden cardiac death is 6 to 9 times greater in the heart failure population, and cardiac arrhythmias are perhaps the leading cause of death in CHF patients. Currently, both the American College of Cardiology and the American Heart Association endorse the placement of implantable cardioverter-defibrillators (ICDs) in patients with ischemic cardiomyopathy, reasonable life expectancy, and reduced ejection fraction below 40% (class I, level of evidence A). Additionally, placement of ICDs is recommended in non-ischemic cardiomyopathy patients who meet similar requirements with an ejection fraction of less than 35% (class I, level of evidence B). Despite these recommendations for primary prevention of sudden death by way of ICD implantation, more than half of the patients receiving a device are likely to not experience an arrhythmic event that necessitates ICD therapy delivery. ICD devices, on average, cost $20,000-50,000 exclusive of operative and follow up costs. Currently, risk stratification of sudden cardiac death and the need for ICD placement are essentially dependent upon assessment of left ventricular ejection fraction. Other methods employed for risk stratification are signal averaged electrocardiogram (ECG) and another electrocardiographic technique known as T-wave alternans. Although these methods are FDA approved for risk prediction of cardiac death, such techniques are not widely employed in the U.S. given equipment and personnel costs to implement them. Thus, alternative testing for risk assessment for the development of sudden cardiac death in the heart failure population is desirable.

Role of Sodium Channels and the SCN5A Gene

The cardiac voltage-gated sodium (Na+) channel, SCN5A, is the main channel generating current for electrical propagation in heart muscle and is the target of many antiarrhythmic drugs. Defective expression of the cardiac Na+ channel results in increased arrhythmic risk as evidenced by sudden death in the Brugada Syndrome. SCN5A mutations have also been implicated in the inherited long-QT syndrome, which can result in the development of the fatal dysrhythmias like ventricular fibrillation and torsades de pointes. Additionally, mutations in the SCN5A gene have also been proposed to exist and enhance risk for drug-induced dysrhythmias.

Many studies have been done to shed light on the role of this tetrodotoxin-insensitive sodium channel in disease states. It has been demonstrated that mutated sodium channels in dilated cardiomyopathy may function differently depending upon the specific mutation type of the principal Na+ channel. Specifically, Nguyen et al have demonstrated that these mutations may lead to changes in physiological function such as slower action potential rise time, enhanced late sodium current during steady state, or impaired inactivation. Additional mutations in the SCN5A gene have been linked to shifts in voltage dependence of Na+ channel inactivation in patients with idiopathic ventricular fibrillation. Prior research has suggested that decreased inactivation of late sodium currents may contribute to action potential prolongation. A different SCN5A gene abnormality has been shown to lead to decreased sodium current density and an positive shift in the cell membrane half-maximal activation potential. Therefore, mutations of the Na+ channel can cause altered channel behavior and arrhythmias.

Previous study showed that disruptions in sodium handling may result in change in calcium homeostasis via action of the Na+/Ca2+ exchanger. Overall, such changes in sodium current (INa) are likely to significantly contribute to arrhythmia in the setting of failing myocardium.

At the genome level, research has focused on the role of SCN5A gene mutations in arrhythmogenesis. Nevertheless, the investigators have recently described acquired defects in Na+ channel messenger RNA (mRNA) that result in reduced Na+ current and occur only in failing hearts. Three 3'-terminal SCN5A mRNA splicing variants were identified and characterized in failing human heart ventricles. Additional measurements suggested that the truncation mutants could cause electrical abnormalities severe enough to contribute to arrhythmic risk. Also, the investigators showed that lymphocytes process sodium channels similarly to cardiomyocytes. Thus, lymphocyte SCN5A mRNA processing may serve as a surrogate marker to assess SCN5A function at the cardiac level and may correlated with arrhythmic risk in high risk populations. This study will determine if SCN5A variant levels are predictive of appropriate ICD therapies in patients with a newly implanted ICD.

ELIGIBILITY:
Inclusion Criteria:

1. All patients must be greater than 18 years of age.
2. All patients must be able to give informed consent.
3. Patients must receive an ICD within 10 days for primary prevention.

Exclusion Criteria:

1. Patients less than 18 years of age.
2. History of congenital heart disease.
3. History of congenital electrophysiological disorders like the long-QT syndrome or Brugada disease.
4. Patients have an ICD implanted for secondary prevention.
5. Patients taking immunosuppressive medications, have chronic infection, or have an acute or chronic inflammatory illness that might alter white cell mRNA expression.
6. Patients with any illness expected to result in death within 18 months of enrollment.
7. Patients with white blood cell dyscrasia or cancers.
8. Patients with end-stage renal disease (ESRD) on hemodialysis or peritoneal dialysis
9. Current illicit drug use.
10. Inability to give informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Estimated)
Dates: Start 2014-06; Primary Completion 2019-07 (Estimated); Study Completion 2020-07 (Estimated)

PRIMARY OUTCOMES:
The levels of sodium channel splicing variants measured by gene expression that are related to arrhythmic events, change every 3 months from baseline to one 1 year after ICD therapy. | baseline, 3-month, 6-month, 9-month, and 12-month after ICD therapy

SECONDARY OUTCOMES:
The levels of sodium channel splicing variants measured by gene expression that are related to the type of ICD implanted, change every 3 months from baseline to one 1 year after ICD therapy. | baseline, 3-month, 6-month, 9-month, and 12-month after ICD therapy

CONTACTS AND LOCATIONS:
Overall Officials: Michael Orlov, MD, Principal Investigator — Rhode Island Hospital
Locations (1):
- Rhode Island Hospital, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hunt SA, Abraham WT, Chin MH, Feldman AM, Francis GS, Ganiats TG, Jessup M, Konstam MA, Mancini DM, Michl K, Oates JA, Rahko PS, Silver MA, Stevenson LW, Yancy CW, Antman EM, Smith SC Jr, Adams CD, Anderson JL, Faxon DP, Fuster V, Halperin JL, Hiratzka LF, Jacobs AK, Nishimura R, Ornato JP, Page RL, Riegel B; American College of Cardiology; American Heart Association Task Force on Practice Guidelines; American College of Chest Physicians; International Society for Heart and Lung Transplantation; Heart Rhythm Society. ACC/AHA 2005 Guideline Update for the Diagnosis and Management of Chronic Heart Failure in the Adult: a report of the American College of Cardiology/American Heart Association Task Force on Practice Guidelines (Writing Committee to Update the 2001 Guidelines for the Evaluation and Management of Heart Failure): developed in collaboration with the American College of Chest Physicians and the International Society for Heart and Lung Transplantation: endorsed by the Heart Rhythm Society. Circulation. 2005 Sep 20;112(12):e154-235. doi: 10.1161/CIRCULATIONAHA.105.167586. Epub 2005 Sep 13. No abstract available. PMID 16160202
- [Background] Rosamond W, Flegal K, Furie K, Go A, Greenlund K, Haase N, Hailpern SM, Ho M, Howard V, Kissela B, Kittner S, Lloyd-Jones D, McDermott M, Meigs J, Moy C, Nichol G, O'Donnell C, Roger V, Sorlie P, Steinberger J, Thom T, Wilson M, Hong Y; American Heart Association Statistics Committee and Stroke Statistics Subcommittee. Heart disease and stroke statistics--2008 update: a report from the American Heart Association Statistics Committee and Stroke Statistics Subcommittee. Circulation. 2008 Jan 29;117(4):e25-146. doi: 10.1161/CIRCULATIONAHA.107.187998. Epub 2007 Dec 17. No abstract available. PMID 18086926
- [Background] Kannel WB, Plehn JF, Cupples LA. Cardiac failure and sudden death in the Framingham Study. Am Heart J. 1988 Apr;115(4):869-75. doi: 10.1016/0002-8703(88)90891-5. PMID 3354416
- [Background] Bardy GH, Lee KL, Mark DB, Poole JE, Packer DL, Boineau R, Domanski M, Troutman C, Anderson J, Johnson G, McNulty SE, Clapp-Channing N, Davidson-Ray LD, Fraulo ES, Fishbein DP, Luceri RM, Ip JH; Sudden Cardiac Death in Heart Failure Trial (SCD-HeFT) Investigators. Amiodarone or an implantable cardioverter-defibrillator for congestive heart failure. N Engl J Med. 2005 Jan 20;352(3):225-37. doi: 10.1056/NEJMoa043399. PMID 15659722
- [Background] Meregalli PG, Wilde AA, Tan HL. Pathophysiological mechanisms of Brugada syndrome: depolarization disorder, repolarization disorder, or more? Cardiovasc Res. 2005 Aug 15;67(3):367-78. doi: 10.1016/j.cardiores.2005.03.005. PMID 15913579
- [Background] Wang Q, Shen J, Splawski I, Atkinson D, Li Z, Robinson JL, Moss AJ, Towbin JA, Keating MT. SCN5A mutations associated with an inherited cardiac arrhythmia, long QT syndrome. Cell. 1995 Mar 10;80(5):805-11. doi: 10.1016/0092-8674(95)90359-3. PMID 7889574
- [Background] Makita N, Horie M, Nakamura T, Ai T, Sasaki K, Yokoi H, Sakurai M, Sakuma I, Otani H, Sawa H, Kitabatake A. Drug-induced long-QT syndrome associated with a subclinical SCN5A mutation. Circulation. 2002 Sep 3;106(10):1269-74. doi: 10.1161/01.cir.0000027139.42087.b6. PMID 12208804